CLINICAL TRIAL: NCT06668480
Title: Effect of Sustained Natural Apophyseal Glide Combined With Strengthening Exercises of Lower Fibers of Trapezius in Patient With Unilateral Neck Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/45
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial having two groups. One group will receive conventional physical therapy along with SNAGS and the second will receive SNAGS and strengthening of lower fibers of trapezius with conventional physical therapy. Both groups will be recruited concurrently.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will not be aware of which group the participant belongs to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SNAGS + Conventional PT Group (Experimental): Participants of this group receive conventional physical therapy.Hot pack and tens ( 10 min each)
  * Sustained natural apophyseal glides to painful or restricted movement
  * 4 sets of 4 repetition per session
  * Strengthening of deep neck flexor
  Interventions: Procedure: Conventional Physical Therapy; Procedure: SNAG'S
- SNAGS+Strengthening of lower fibers trapezius+Conventional PT Group (Experimental): * Participants of this group receive conventional physical therapy. It will comprise of hot pack for 10 minutes, TENs at 80-100 Hz over trapezius for 10 minutes.
  * Sustained natural apophyseal glides to painful or restricted movement.4 sets of 3-5 repetition per session.
  * Strengthening of deep neck flexors
  * Then strengthening exercises of lower fibers of trapezius
  Interventions: Procedure: Conventional Physical Therapy; Procedure: Strengthening Exercise; Procedure: SNAG'S

INTERVENTIONS:
Procedure: Conventional Physical Therapy — It will comprise of hot pack for 10 minutes, TENs at 80-100 Hz over trapezius for 10 minutes.Strengthening of deep neck flexors
Procedure: Strengthening Exercise — Strengthening exercises of lower fibers of trapezius
  Arms: SNAGS+Strengthening of lower fibers trapezius+Conventional PT Group
Procedure: SNAG'S — Sustained natural apophysial glides will consist of frequency: 4 sets of 3-5 repetition per session for 2 weeks

SUMMARY:
Neck pain is considered one of the very common cause behind musculoskeletal pain and is 4th leading cause of disability . Cervical pain is among 5 most contributing factors in causing years lived with disability.Individuals with unilateral neck pain exhibit significantly less Lower Trapezius strength than Middle and Upper Trapezius fibers .Mulligan is one of the mobilization techniques that can be applied in case of neck pain.In prolong neck pain there is a hyperactivation and shortening of upper trapezius which makes the lower trapezius weak this leads to imbalance between cervical and scapular muscles and result in impaired biomechanics. So mostly treatment focused on upper trapezius and neglecting the lower trapezius and this create increase chances of recurrency of neck pain because the imbalance remains present. So, this study aims at evaluating the effects of SNAGS combined with strengthening exercises of lower fibers of trapezius .

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-35 years
* Both gender
* Unilateral neck pain
* Symptoms of duration more than 3 months.
* NPRS scoring of greater than or equal to 4 points.
* Neck disability index score of 20% or above.
* Manual muscle testing : grade 3

Exclusion Criteria:

* Prior cervical and thoracic spine fractures, dislocations, or surgeries, spinal osteoporosis or infection, or whiplash.
* Any trauma or localized infection in neck region
* Psychiatric diseases such as phobia/obsession and depression

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 2 weeks
  Pain will be measured on the basis of Numeric Pain Rating Scale score.It is rated on 0-10 scale in which 0 means no pain and 10 means the maximum possible pain
ROM | 2 weeks
  Cervical ROM will be measured through CROM device
Level of Neck Disability | 2 weeks
  Neck Disability Index will be used to measure level of neck disability
Muscle strength | 2 weeks
  MMT for Lower fibers of trapezius

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan